CLINICAL TRIAL: NCT03630692
Title: Safety and Compliance of Patients Treated With Oral Route Anti Cancer Drugs.
Brief Title: Safety and Compliance of Renal Cancer Patients Treated by Non-IV Drugs
Acronym: TOPTACOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: University of Angers, GRANEM (Unknown); Fondation ARC (Other)
Responsible Party: Sponsor
Other Study IDs: TOPTACOS
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Renal Cancer; Stage III Renal Cell Cancer
Keywords: kidney cancer,; oral drug; safety; adherence
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observance of oral drug treatment: Study of observant or nonobservant patient behavior for their oral drug treatment
  Interventions: Drug: observance of oral drug treatment

INTERVENTIONS:
Drug: observance of oral drug treatment — Completion of questionnaires at 4 times during patient's oral route drug treatment
  Other Names: oral drug treatment

SUMMARY:
Generally, in the trials, an observant patient is described as correctly taking 90 to 100% of the prescribed doses. Here, the 80% compliance rate will be the cut-off between observant and non-observant patients.

The evaluation methodology is based primarily on a survey of patients with metastatic or locally advanced kidney cancer who have just began an oral treatment protocol. The constitution of this cohort will be made from newly treated patients included by oncologists. The survey consists of implementing a series of questionnaires with each patient of the sample throughout the course of oral cancer care.

This series of questionnaires will aim to identify:

* the gradient of compliance of the patient with his treatment,
* all the factors likely to influence positively or negatively the latter, whether medical, material or socio-economic,
* the evolution of patient compliance during their treatment course,
* a patient's quality of life index through the standardized quality of life survey form (EORTC - Quality of Life Questionnaire QLQ C30 version 3).
* These questionnaires will be supplemented by the medical record data (including information on tolerance and possible drug interactions). The representativeness of the patients surveyed will be established by comparing the statistical characteristics of the surveyed population with those of the aggregate anonymous global data obtained by the two Medical Department of the French Regional Health Insurance of the two regions. From the data compiled by this study, different econometric models of patient behavior will seek to establish, in particular, a relationship between the probability that a given patient will be either non or poorly observant and the various variables proved to be statistically significant.

DETAILED DESCRIPTION:
Data obtained from patients via the questionnaires will be copied into a computer database and as follows :

* The date of birth (day, month and year),
* Sex,
* The patient's opinion and attitude towards the current treatment: compliance, adverse effects, lifestyle restrictions, changes in professional activity, family activities, relationships, physical fitness, moral, concomitant treatments, expenses not refunded parallels related to the management of adverse effects,
* The family situation, the number of children,
* Degrees obtained and employment,
* Net monthly income.

In parallel with the questionnaires, the Clinical Research Associate (CRAs) of the Observatory will collect data from the medical file on site. The data collected on an electronic Case Report Form (e-CRF) are as follows:

* Type of cancer, date of diagnosis and metastatic disease, possible surgery and radiotherapy,
* Description of the different treatment lines: number of cures, start and end date, response, toxicities,
* Status of the patient at the end of the study.

The number of subjects needed is calculated from observant patients. Based on the existing literature on adherence to chemotherapy or targeted oral therapy, the observed compliance rate is approximately 80%. However, since this characteristic is the object of this study and therefore not known ex ante, in the calculations of the sample size, the value allowing to obtain the lowest margin of error on the rate of compliance, an estimated prevalence of 50% compliance is used. By setting the risk of the first species at 5%, a confidence level of 95%, it is then necessary to include 132 patients.

In addition, given the difficulty inherent in the questionnaires in collecting all the information, 20% of the data was estimated not to be evaluable. It will therefore be necessary to include 158 patients in the study to reach our goal.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with metastatic or locally advanced kidney cancer
* Patient initiating for the first time an oral route anticancer drug : Sutent® (sunitinib), Nexavar® (sorafenib), Afinitor® (everolimus), Votrient® (pazopanib) and Inlyta® (axitinib) and Cabometyx® (cabozantinib)
* Patient having signed an informed consent
* Patient treated outside interventional clinical trial

Exclusion Criteria:

* Patient with cancer other than kidney cancer
* Patient with non-extensive kidney cancer
* Patient treated by surgery, radiotherapy and intravenous chemotherapy exclusively
* Patient unable to undergo protocol monitoring
* Patient included in an interventional trial
* Patient refusing a survey at home or having hearing problems
* Other medical conditions that may interfere with the understanding of the informed consent document, with the assessment of tolerance and the response to questionnaires
* Patient with another condition deemed incompatible with the patient's inclusion into the protocol.
* Patient under guardianship or trusteeship, deprived of liberty, underage patient or pregnant woman
* Patient not affiliated with a social security system beneficiary of such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for a metastatic renal cancer by an oral route drug (sunitinib, axitinib, sorafenib, pazopanib, everolimus et cabozantinib) in Bretagne and Pays de la Loire area
Sampling Method: Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2016-03-25 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Study of observant or nonobservant patient behavior via patient questionnaire | 11 months
  Observance is first calculated via the use of the Morisky's score. The value of the score is between 0 and 4. The 0 corresponds to the absence of observance, the 4 to the perfect observance.
  This score is completed by a question about drug delay (which measures poor compliance).
  A subjective measure of compliance is also obtained from the patient's positioning of his compliance on a scale from 0 to 10. The value 0 corresponds to the fact that the person indicates that they do not comply at all with the treatment prescribed by the oncologist. Conversely, the value 10 corresponds to the exact respect of the treatment prescribed by the oncologist.
  These two indicators are measured at different periods of treatment (1 month, 4 months ; 7 months and 10 months) via a patient questionnaire.

SECONDARY OUTCOMES:
Oral route Progression Free Survival evaluation (PFS) | 11 months
  PFS (duration between treatment start and progression date) will be evaluated via medical records analysis.
Oral route Response rate analysis | 11 months
  Response rate will be evaluated via medical records analysis.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | 11 months
  adverse event due to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francoise GRUDE, Pharmacist, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (14):
- France (14):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU, Angers
  - Clinique Pasteur Saint Esprit, Brest
  - CHU Morvan, Brest
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier, Le Mans
  - Clinique Victor Hugo, Le Mans
  - Centre Catherine de Sienne, Nantes
  - CHIC Quimper, Quimper
  - Centre Eugène Marquis, Rennes
  - CHP, Saint-Grégoire
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Hospitalier, St-Malo
  - CHP Océane, Vannes